CLINICAL TRIAL: NCT04020900
Title: Respiratory Management of Children Under Anaesthesia: a French Prospective Multicentre Observational Study
Brief Title: Respiratory Management of Children Under Anaesthesia
Acronym: PEDIAVENT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Pediavent
Record Dates: First submitted 2019-07-15; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia; Peroperative Complication
Keywords: Children; Respiratory
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children <18 years, admitted for a general anesthesia.: Children <18 years, admitted for a general anesthesia.
  Interventions: Other: Respiratory management

INTERVENTIONS:
Other: Respiratory management — Data on respiratory management were collected at different time: data regarding the induction period, ventilatory parameters set and measured during a stable period, ventilatory change made during anaesthesia, use of recruitment manoeuvres, data regarding weaning and extubation

SUMMARY:
Ventilation management in paediatric anaesthesia remains difficult because of the wide range of age and weight, and therefore practices are heterogeneous. In adults, protective ventilation during anesthesia is now a standard of care but in children there is no level of evidence to recommend it. The aim of the study was to describe current practice and the factors associated with the use of high tidal volume during anaesthesia in children in France.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years of age
* Admitted in one of the participating centers
* over 2 days (21 and 22 June 2017)

Exclusion Criteria:

* Children extracorporeal circulation
* Children who required ventilation with lung exclusion
* Opposition of the parents or legal guardians

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children < 18 years of age, admitted for a general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving a tidal volume higher than 10 milliliters/kilogram (ml/kg) of actual body weight | up to 1 hour (during a stable period in anaesthesia)
  Number of patients receiving a tidal volume higher than 10 milliliters/kilogram (ml/kg) of actual body weight

CONTACTS AND LOCATIONS:
Overall Officials: Florent BAUDIN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France